CLINICAL TRIAL: NCT05842928
Title: Patient-centred Deprescribing of Psychotropic, Sedative and Anticholinergic Medication in Elderly Patients With Polypharmacy: a Cluster-randomised Trial
Brief Title: Patient-centred Deprescribing of Psychotropic, Sedative and Anticholinergic Medication in Elderly Patients With Polypharmacy
Acronym: PARTNER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Bielefeld University (Other); University of Witten/Herdecke (Other); University Hospital Heidelberg (Other); University Hospital Regensburg (Other); Institute for Applied Quality Improvement and Research in Health Care (Unknown); Techniker Krankenkasse (Other); Federal Joint Committee (Other Government)
Responsible Party: Principal Investigator, Tobias Dreischulte, Professor of Clinical Health Services Research, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 01VSF21038
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Deprescriptions; Antidepressive Agents; Antipsychotic Agents; Analgesics, Opioid; Hypnotics and Sedatives; Cholinergic Antagonists
Keywords: Polypharmacy; General Practice; Primary Health Care; Pharmacies; Medication Safety

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: To avoid selection bias and Hawthorne bias, the collaborating units (GP practice and community pharmacy) in the intervention group are blinded to the target drugs (PSA-PIM) until the time of randomisation, and in the control group until the end of the study. The same applies to patient participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Intensified and patient-centred cooperation between GPs and pharmacists including patient empowerment
  Interventions: Behavioral: PARTNER intervention
- Control Arm (Active Comparator): Extended routine care
  Interventions: Behavioral: Control intervention

INTERVENTIONS:
Behavioral: PARTNER intervention — The PARTNER intervention includes the following components:
  1. Education for health care professionals
     A) written manual on deprescribing PSA-PIM, which consists of brief information and more detailed explanations;
     B) access to digital instructional videos/podcasts that address potential problems in deprescribing and provide possible solutions;
     C) checklist for identification of drug-related problems for pharmacists;
     D) tapering support tool to facilitate the selection of tapering schemes;
     E) divisibility list for PSA-PIM to support the implementation of tapering schemes;
     F) empowerment brochures for patients each focussing on one PSA-PIM subgroup
  2. Interprofessional workshop and case conference for GPs and pharmacists
  3. Pharmacy visit (brown bag/medication review) including patient empowerment
  4. GP practice visit including shared decision making (SDM)
  Arms: Intervention Arm
Behavioral: Control intervention — The control intervention only comprises a pharmacy visit with brown bag review.
  Arms: Control Arm

SUMMARY:
The PARTNER study is a multicentre, two-arm, pragmatic cluster-randomised trial evaluating the impact of a focused and patient-centred cooperation between general practitioners (GPs) and community pharmacists (PARTNER intervention) on reductions in the use of psychotropic, sedative and anticholinergic potentially inappropriate medication (PSA-PIM) compared to a control intervention. The PARTNER intervention comprises (1) education for health care professionals, (2) an interprofessional workshop and case conference, (3) a pharmacy visit with brown bag/medication review and patient empowerment, (4) GP practice visit with shared decision making. The control intervention only comprises a pharmacy visit with brown bag review.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older
* Patient is capable of giving consent
* GP contact in the quarter prior to inclusion
* Current use of ≥ 5 drugs, including ≥ 1 PSA-PIM (hypnotics, opioids, gabapentinoids, antipsychotics, antidepressants, anticholinergic urospasmolytics) with a treatment duration of ≥ 6 months
* Willingness to select a regular pharmacy for the study period
* Consent to data exchange between GP and community pharmacy

Exclusion Criteria:

* Terminal illness (life expectancy < 6 months)
* Current treatment of pain associated with cancer
* Other serious physical illness or mental distress (e.g. bereavement) that makes participation in the study impossible (according to the GP's assessment)
* Psychiatric illness or addiction that makes participation in the study impossible (according to the GP's assessment)
* Unable to meet the requirements of the study (participation in telephone or written questionnaires, visits to the GP practice or community pharmacy, alone or with the help of caregivers for physical infirmity)
* Current participation in research projects on medication safety or geriatric medicine

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2023-03-25 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Reduction in the PSA-PIM Drug Burden Index (DBI) by ≥ 0.15 points | 6 months
  Clinically relevant reduction in PSA-PIM exposure at patient level after 6 months follow-up, as measured by the Drug Burden Index method. The primary endpoint is defined as a responder endpoint at patient level, where response is defined as a reduction in the Drug Burden Index (DBI) by ≥ 0.15 points (Primary endpoint: T2 vs T0)

SECONDARY OUTCOMES:
Reduction in the PSA-PIM Drug Burden Index (DBI) by ≥ 0.15 points | 12 months
  Clinically relevant reduction in PSA-PIM exposure at patient level after 12 months follow-up, as measured by the Drug Burden Index method (T4 vs T0)
Frequency of deprescribing PSA-PIM stratified by PSA-PIM subgroups | 12 months
  Proportion (%) of patients with a reduction in DBI ≥ 0.15 (T2 vs T0; T4 vs T0)
Total exposure with PSA-PIM | 12 months
  Average of the Drug Burden Index (DBI); mean change in the number of PSA-PIM taken (T2 vs T0; T4 vs T0)
Total exposure to PSA-PIM stratified by PSA-PIM subgroups | 12 months
  Average of the Drug Burden Index (DBI); mean change in the number of PSA-PIM taken (T2 vs T0; T4 vs T0)
Frequency of new PSA-PIM prescriptions | 12 months
  Proportion (%) of patients with a new prescription of ≥1 PSA-PIM (T2 vs T0; T4 vs T0)
Frequency of taking other potentially inappropriate medication (PIM) (Validated PIM lists, e.g. PRISCUS list, START/STOPP, Anticholinergic Burden) | 12 months
  Average change in the number of PIMs (T2 vs T0; T4 vs T0)
Number of falls and hospitalisations due to fall events (Falls diary, Hospitalisation diary according to FIMA) | 12 months
  Proportion (%) of patients with falls/hospitalisations due to fall injuries (T2 vs T0; T4 vs T0)
Cognition (Verbal Fluency Test) | 12 months
  Average (T2 vs T0; T4 vs T0)
Quality of life (EQ5-D-5L) | 12 months
  Average (T2 vs T0; T4 vs T0)
Insomnia (Regensburg Insomnia Scale; RIS) | 12 months
  Change from baseline in psychological symptoms and sleep assessed with the Regensburg Insomnia Scale (RIS). RIS includes 10 questions on cognitive, emotional and psychophysiological aspects of a sleep disorder. Five answer options for each question are possible (scored 0 to 4; higher scores indicate higher burden). The overall RIS score is the sum of the scores from each of the 10 questions. The overall RIS score can therefore range from zero to 40.
  Average (T2 vs T0; T4 vs T0)
Adverse drug reactions (ADRs) | 12 months
  Average (T2 vs T0; T4 vs T0)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Dreischulte, Prof. Dr., Principal Investigator — Institute of General Practice and Family Medicine, University Hospital, LMU Munich, Munich, Germany
Locations (3):
- Germany (3):
  - University of Bielefeld, Bielefeld
  - University Hospital, LMU Munich, Munich
  - Witten/Herdecke University, Witten

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haerdtlein A, Bernartz K, Peter S, Lepenies LK, Puzhko S, Eberhardt Y, Maas M, Picker-Huchzermeyer S, Brisnik V, Falomir D, Gensichen J, Steimle T, Huppertz G, Koller M, Zeman F, Vanella P, Seidling HM, Mortsiefer A, Muth C, Dreischulte T. General practitioner-pharmacist collaboration to enhance deprescribing of psychotropics, sedatives, and anticholinergics among older polypharmacy patients in primary care: study protocol of a cluster-randomized controlled trial (PARTNER). Ther Adv Drug Saf. 2026 Jan 8;17:20420986251400042. doi: 10.1177/20420986251400042. eCollection 2026. PMID 41522713